CLINICAL TRIAL: NCT03078517
Title: Comparison of the LMA Protector and the I-gel in Anesthetized Patients.
Brief Title: Comparison of the LMA Protector and the I-gel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Associate professor, SMG-SNU Boramae Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20170104
Record Dates: First submitted 2017-01-04; First posted 2017-03-13 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Mechanical Ventilation
Keywords: I-gel; Laryngeal mask airway protector

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-gel group (Active Comparator): After the induction of anesthesia, I-gel is inserted into the oropharyngeal space.
  Interventions: Device: I-gel
- LMA protector group (Experimental): After the induction of anesthesia, laryngeal mask airway protector is inserted into the oropharyngeal space.
  Interventions: Device: Laryngeal mask airway protector

INTERVENTIONS:
Device: I-gel — After the induction of anesthesia, i-gel is inserted along the palatopharyngeal curve.
  Arms: I-gel group
Device: Laryngeal mask airway protector — After the inudction of anesthesia, laryngeal mask airway protector is inserted along the palatopharyngeal curve, and the cuff is inflated.
  Arms: LMA protector group

SUMMARY:
Investigators aim to compare two supraglottic airway devices; the i-gel and the newly developed laryngeal mask airway protector in terms of airway sealing effect, the insertion success rate, and the incidence of complications in anesthetized patients.

ELIGIBILITY:
Inclusion Criteria:

* Requirement for mechanical ventilation under general anesthesia

Exclusion Criteria:

* Surgical position other than supine position
* Tumors or anatomical abnormalities in the upper airway
* Known or predicted difficult airway
* Body mass index > 30 kg/m2
* Required postoperative mechanical ventilation
* Head and neck surgery
* Aspiration tendency

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2018-01-20 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal airway leak pressure | At 5 min after the insertion of i-gel or LMA protector
  Oropharyngeal airway leak pressure is measured by closing the expiratory valve of the circle system at a fresh gas flow of 3 L/min and observing the airway pressure at equilibrium.

SECONDARY OUTCOMES:
Number of insertion attempt for the successful placement | During the insertion of i-gel or LMA protector
  The numbers of insertion attempt for successful placement are counted.
Insertion time | During the insertion of i-gel or LMA protector
  Insertion time is defined as the time from picking up the device to confirming successful placement (the appearance of the ETCO2 on the monitor screen).
Ease of insertion | During the insertion of i-gel or LMA protector
  Ease of insertion is defined as follows. Easy: requiring no additional maneuver, fair: requiring 1 additional maneuver, difficult: requiring more than 1 additional maneuver.
Ease of gastric tube insertion | At 25 min after the insertion of i-gel or LMA protector
  Ease of garstic tube insertion is assessed as follows; easy, difficult, impossible.
The accuracy of insertion location of the device in the oropharyngeal space | At 15 min after the insertion of i-gel or LMA protector
  After insertion of the device, the insertion location is assessed using a fiberoptic bronchoscope; 4, only the vocal cords seen; 3, vocal cords and posterior part of the epiglottis seen; 2, vocal cords and anterior part of the epiglottis seen; 1, vocal cords not seen, but adequate ventilation.
Blood staining on the i-gel or LMA protector | Immediately after removal of i-gel or LMA protector
  After removal of the device, the presence of blood staining on the device is checked.
The incidence and severity of postoperative sore throat | At 1 and 24 h after surgery
  Postoperative sore throat is assessed using a numerical rating scale (0-100 point).

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Young Hwang, M.D., Ph.D., Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang JE, Kim H, Lee JM, Min SW, Won D, Jun K, Hwang JY. A prospective, randomized comparison of the LMA-protector and i-gel in paralyzed, anesthetized patients. BMC Anesthesiol. 2019 Jul 4;19(1):118. doi: 10.1186/s12871-019-0785-8. PMID 31272379